CLINICAL TRIAL: NCT00918385
Title: A Phase II Trial of Genomic Guided Therapy With Dasatinib or Nilutamide in Metastatic Castration-Resistant Prostate Cancer
Brief Title: Genomic Guided Therapy With Dasatinib or Nilutamide in Metastatic Castration-Resistant Prostate Cancer
Acronym: ARS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Permanent closure of trial to further accrual based on IDE disapproval
Sponsor: Duke University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00012159; CA180-263
Record Dates: First submitted 2009-06-10; First posted 2009-06-11 (Estimated); Results first posted 2014-10-29 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-09

CONDITIONS: Prostate Cancer
Keywords: hormone resistant prostate cancer; castration resistant prostate cancer; hormone refractory prostate cancer; metastatic prostate cancer; hormonal therapy; antiandrogen therapy; androgen receptor; nilutamide; dasatinib; genomics; genomic signature; genomic predictor; genomic analysis; genomic expression profile
MeSH Terms: conditions — Prostatic Neoplasms; Bulbo-Spinal Atrophy, X-Linked | interventions — nilutamide; Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): High Androgen Receptor (AR) activity
  Interventions: Drug: Nilutamide
- 2 (Active Comparator): Low Androgen Receptor (AR) activity
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Nilutamide — Nilutamide 150mg orally each day for 28 days per cycle. After first progression, Nilutamide 150mg orally each day in combination with Dasatinib 100mg orally each day for 28 days per cycle.
  Other Names: Nilandron
  Arms: 1
Drug: Dasatinib — Dasatinib 100mg orally daily x 28 days per cycle. After first progression, Dasatinib 100mg orally each day in combination with Nilutamide 150mg orally each day for 28 days per cycle.
  Other Names: Sprycel
  Arms: 2

SUMMARY:
This is a phase II multi-center study to determine the clinical impact of using a patient-specific genomic expression signature of androgen receptor (AR) activity to determine therapy for patients with castration-resistant metastatic prostate cancer (CRPC). After patient eligibility is determined, the genomic signature will be applied to fresh frozen tissue harvested from a metastatic lesion during image-guided biopsy. After assessing for androgen receptor activity, the investigators will select patients for either continued androgen manipulation with nilutamide (high AR activity) or targeted therapy with dasatinib (low AR activity). Once patients develop a first progression on either arm, patients will receive combination therapy with dasatinib and nilutamide. The primary aim is to estimate the median progression free survival in men with CRPC treated according to tumor AR activity. The investigators hypothesize that by treating men based upon AR activity, median progression free survival (PFS) will improve from a historical median of 3.0 months to 6.0 months.

DETAILED DESCRIPTION:
Prostate cancer is the most commonly diagnosed non-cutaneous malignancy of men in the United States and remains the second leading cause of cancer-related mortality among men. Novel approaches are necessary to personalize and improve treatment. The androgen receptor (AR) plays a critical role in the normal development and function of the prostate and promotes growth in most prostate cancers. Most patients with advanced prostate cancer have cancer that will initially respond to androgen-targeting therapy (focusing on decreasing the circulating levels of testosterone which is the primary source of ligand for the AR receptor). However, castrate resistance usually develops within 18 to 24 months and the median survival of men with castration resistant prostate cancer (CRPC) ranges between 12 to 18 months. Current options are limited including: secondary hormonal manipulations, radiopharmaceuticals, and chemotherapy and only docetaxel, a taxane that targets microtubules, has been proven to prolong survival.

Importantly, it has become clear that for some patients with CRPC, the prostate tumors remain dependent on AR activity. This has been supported by studies demonstrating different genetic and metabolic mechanisms by which prostate cancer cells maintain AR activity despite low levels of circulating androgen. An assay detecting AR activity that more comprehensively reflects the variety of mechanisms by which AR activity is preserved has the potential to accurately differentiate between men who have tumors still dependent on AR activity from those that are truly independent of AR activity. The identification of patients with continued AR activity has the potential to improve response to secondary hormonal manipulations; men with tumors having low levels of AR activity are likely to require alternative approaches.

We have developed a transcriptional "signature" for AR activity with the goal of identifying the true status of AR in tumors of men with CRPC. After validating the AR signature on in vitro and human prostate samples to ensure that it accurately and reproducibly detects AR activity, we applied the AR signature to several independent datasets to determine the distribution of CRPC tumors with preserved AR activity. Interestingly, there is consistent heterogeneity with respect to predicted AR activity. While overall AR activity decreases in CRPC, there is a subgroup of patients with persistently elevated AR activity. In tumors with low AR activity, we observed that the probability of AR activity was negatively correlated with predicted SRC activity in localized prostate cancer and CRPC.

Patients with persistently high AR activity will be treated with nilutamide, an approved oral agent used in metastatic CRPC to target the AR. Patients with tumors having low AR activity will be treated with dasatinib (an oral drug known to target the SRC family kinases). As there is compelling pre-clinical evidence of interactions between the SRC pathway and AR signaling, patients failing either single agent treatment will be treated with the combination of nilutamide and dasatinib and followed again for progression.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of adenocarcinoma of the prostate.
2. Radiographic evidence of metastatic disease amenable to image-guided biopsy.
3. Testosterone <50ng/dL on androgen deprivation therapy (ADT). ADT must continue while on study.
4. The patient must have discontinued antiandrogens 30 days prior to baseline PSA unless the patient did not respond to anti-androgen therapy or experienced a decline in PSA lasting < 3 months after starting antiandrogen therapy.
5. Evidence of disease progression on ADT.
6. Patients must have adequate organ and marrow function as defined below:

   * Hemoglobin >9.0g/dL (without transfusion of PRBC)
   * ANC/AGC >1,500/μl
   * Platelets >75,000/μl
   * Total bilirubin < 2.0 times the institutional ULN
   * Creatinine <1.5 times the institutional ULN
   * PT or INR and aPTT < 1.5 times the institutional ULN
   * AST and ALT <2.5 x ULN
7. Age > 18 years
8. Ability to take oral medications (pills must be swallowed whole)
9. ECOG performance status 0-2
10. Concomitant Medications:

    * Patient agrees to discontinue and not to initiate taking St. Johns Wort while receiving dasatinib therapy (discontinue St. Johns Wort at least 5 days before starting dasatinib)
    * Patient agrees not to initiate IV bisphosphonates while on dasatinib. Patients on IV bisphosphonates for > 4 weeks prior to dasatinib will continue on therapy
11. Men of reproductive potential who have not had a radical prostatectomy must agree to use an effective contraceptive method. Patients who have had a prostatectomy are sterile and do not need to use contraception
12. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

1. Patients who have received prior treatment with nilutamide or dasatinib
2. Patients who have not recovered to Grade 1 or Grade 0 from the toxic effects of prior investigational therapy, biologic therapy, hormonal therapy (other than ADT), immunotherapy, or chemotherapy
3. Medical contraindications to stopping aspirin or coumadin for 1 week prior to image-guided tumor biopsy AND while on dasatinib treatment.
4. History of the following cardiac related conditions:

   * Uncontrolled angina, congestive heart failure or MI within (6 months)
   * Diagnosed congenital long QT syndrome
   * Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes)
   * Prolonged QTc interval on pre-entry electrocardiogram (> 450 msec)
   * Subjects with hypokalemia or hypomagnesemia if it cannot be corrected prior to dasatinib administration
5. History of significant bleeding disorder unrelated to cancer.
6. Concomitant use of Category I drugs that are generally accepted to have a risk of causing Torsades de Pointes including: (These medications can be stopped while the patient is on the protocol and the patient needs to be off the drugs for at least 7 days prior to starting dasatinib)
7. Patients who have a history of amiodarone use.
8. Clinically significant pericardial or pleural effusion or severe respiratory insufficiency
9. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (requiring antifungal, antibiotic or antiviral therapy), symptomatic congestive heart failure (NYHC II or greater, unstable angina pectoris, cardiac arrhythmia (uncontrolled SVT or any VT), or psychiatric illness/social situations that would limit compliance with study requirements.
10. Patients with a medical contraindication to image-guided biopsies

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2009-05; Primary Completion 2012-02 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel George, MD, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - University of Washington/Seattle Cancer Care Alliance, Seattle, Washington

REFERENCES:
- [Background] Mendiratta P, Mostaghel E, Guinney J, Tewari AK, Porrello A, Barry WT, Nelson PS, Febbo PG. Genomic strategy for targeting therapy in castration-resistant prostate cancer. J Clin Oncol. 2009 Apr 20;27(12):2022-9. doi: 10.1200/JCO.2008.17.2882. Epub 2009 Mar 16. PMID 19289629

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Accrual open from January 2009 to July 2011 in these institutions: Dana Farber Cancer Institute, Duke Cancer Institute, MD Anderson Cancer Center, Oregon Health & Science Univ, U of CA at San Francisco, U of Washington.
Pre-assignment Details: 64 consented, 7 screen failures. Of the 57 who began enrollment, 2 not assigned to treatment (withdrew consent, clinically unstable), 22 QC technical failures (received dasatinib off study) and 33 assigned per protocol (15 high AR, 18 low AR), 2 progressed before treatment. 14 high AR and 17 low AR began treatment and are included in the analysis.
Groups:
- Arm 1=High AR Nilutamide: High Androgen Receptor (AR) activity of >= 0.50
  Nilutamide: Nilutamide 150mg orally each day for 28 days per cycle. After first progression, Nilutamide 150mg orally each day in combination with Dasatinib 100mg orally each day for 28 days per cycle.
- Arm 2= Low AR Dasatinib: Low Androgen Receptor (AR) activity of < 0.50
  Dasatinib: Dasatinib 100mg orally daily x 28 days per cycle. After first progression, Dasatinib 100mg orally each day in combination with Nilutamide 150mg orally each day for 28 days per cycle.
Period: Monotherapy
Arm/Group | Arm 1=High AR Nilutamide | Arm 2= Low AR Dasatinib
Started | 14 | 17
Completed | 12 (Completed = received treatment until first disease progression on single agent.) | 11 (Completed = received treatment until first disease progression on single agent.)
Not Completed | 2 | 6
Not completed — Adverse Event | 1 | 6
Not completed — Complicating illness | 1 | 0
Period: Combination Nilutamide and Dasatinib
Arm/Group | Arm 1=High AR Nilutamide | Arm 2= Low AR Dasatinib
Started | 12 | 11
Completed | 6 | 3
Not Completed | 6 | 8
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Complicating illness | 1 | 0
Not completed — Withdrawal by Subject | 2 | 7

BASELINE CHARACTERISTICS:
Population: 64 consented but 7 screen failures, so 57 enrolled. 2 never assigned to rx (withdrew consent, clinically unstable), 33 assigned by AR activity (15 high AR to nilutamide, 18 low AR to dasatinib) and 22 QC technical failures (received dasatinib). 14 of 15 high AR and 17 of 18 low AR began protocol treatment. Analyses include the 31 treated patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1=High AR Nilutamide | Arm 2= Low AR Dasatinib | Total
Number analyzed (Participants) | 14 | 17 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 4 | 10
  >=65 years | 8 | 13 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 14 | 17 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 13 | 15 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 17 | 31

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is the interval from start of monotherapy until first disease progression or death, whichever occurred first.
Time Frame: During monotherapy ( at least 12 weeks)
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Arm 1=High AR Nilutamide | Arm 2= Low AR Dasatinib
Number analyzed (Participants) | 14 | 17
months | 2.8 [2.7 to 4.4] | 2.6 [1.1 to 3.0]

2. Secondary Outcome: Overall Response Rate of Men With High AR Activity
Description: Tumor response was based on Response Criteria in Solid Tumors (RECIST). Complete response (CR) is defined as disappearance of all target and non-target lesions and normalization of tumor marker level. Partial response (PR) is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Time Frame: During monotherapy (at least 12 weeks)
Population: 14 subjects began treatment; 13 with response documentation are included in the calculation; 1 subject was omitted because response documentation was not provided.
Measure: Number (95% Confidence Interval); unit: percentage of patients with CR,PR
Arm/Group | Arm 1=High AR Nilutamide
Number analyzed (Participants) | 13
percentage of patients with CR,PR | 0 [0 to 23]

3. Secondary Outcome: Overall Response Rate of Men With Low AR Activity
Description: Tumor response is based on Response Evaluation Criteria in Solid Tumors (RECIST). Complete response (CR) is defined as disappearance of all target and non-target lesions and normalization of tumor marker level. Partial response (PR) is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Time Frame: During dasatinib monotherapy ( at least 12 weeks)
Population: Of the 17 subjects treated, 15 had response documentation and are included in the calculation. Two were omitted (1 because response documentation was not provided; 1 ended treatment after 2 weeks for toxicity prior to repeat scans).
Measure: Number (95% Confidence Interval); unit: percentage of patients with CR,PR
Arm/Group | Arm 2= Low AR Dasatinib
Number analyzed (Participants) | 15
percentage of patients with CR,PR | 0 [0 to 21]

ADVERSE EVENTS:
Arm/Group | Arm 1=High AR Nilutamide | Arm 2= Low AR Dasatinib | Combination Nilutamide and Dasatinib
Serious Adverse Events (participants affected / at risk) | 14/14 | 16/17 | 14/23
Other Adverse Events (participants affected / at risk) | 3/14 | 1/17 | 1/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1=High AR Nilutamide (N=14) | Arm 2= Low AR Dasatinib (N=17) | Combination Nilutamide and Dasatinib (N=23)
Anemia (Blood and lymphatic system disorders) | 11 | 11 | 13
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | 0
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0
Blurred vision (Eye disorders) | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 1
Eye disorders - Other (Eye disorders) | 9 | 0 | 5
Eye pain (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 1
Anal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 4 | 6 | 7
Diarrhea (Gastrointestinal disorders) | 4 | 4 | 4
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Fecal incontinence (Gastrointestinal disorders) | 2 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 2 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 | 1 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 10 | 6 | 7
Rectal pain (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 3 | 2
Edema limbs (General disorders) | 4 | 4 | 1
Edema trunk (General disorders) | 1 | 1 | 0
Fatigue (General disorders) | 4 | 11 | 10
Fever (General disorders) | 1 | 1 | 0
Flu like symptoms (General disorders) | 1 | 0 | 1
Pain (General disorders) | 6 | 4 | 2
Gum infection (Infections and infestations) | 1 | 0 | 0
Infections and infestations - Other (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1
Creatinine increased (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 4 | 0
Platelet count decreased (Investigations) | 1 | 3 | 2
Weight loss (Investigations) | 0 | 1 | 3
White blood cell decreased (Investigations) | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 3 | 7 | 6
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 5 | 4
Ataxia (Nervous system disorders) | 0 | 1 | 0
Cognitive disturbance (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 2 | 2
Dysgeusia (Nervous system disorders) | 0 | 3 | 0
Headache (Nervous system disorders) | 2 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 3 | 3
Sinus pain (Nervous system disorders) | 0 | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 2
Depression (Psychiatric disorders) | 2 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 2 | 2
Hematuria (Renal and urinary disorders) | 1 | 2 | 1
Renal and urinary disorders - Other (Renal and urinary disorders) | 2 | 1 | 1
Urinary frequency (Renal and urinary disorders) | 1 | 1 | 2
Urinary incontinence (Renal and urinary disorders) | 2 | 0 | 0
Urinary retention (Renal and urinary disorders) | 2 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0
Urine discoloration (Renal and urinary disorders) | 0 | 1 | 0
Gynecomastia (Reproductive system and breast disorders) | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 2 | 2 | 3
Scrotal pain (Reproductive system and breast disorders) | 1 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 4
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 1 | 0
Hot flashes (Vascular disorders) | 4 | 1 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0
Extraocular muscle paresis (Eye disorders) | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Rhinitis infective (Infections and infestations) | 0 | 0 | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 0 | 2
Dysgeusia (Nervous system disorders) | 0 | 0 | 5
Headache (Nervous system disorders) | 0 | 0 | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1=High AR Nilutamide (N=14) | Arm 2= Low AR Dasatinib (N=17) | Combination Nilutamide and Dasatinib (N=23)
Anemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Obstruction, GU:Ureter (Renal and urinary disorders) | 1 | 0 | 0
Eye disorders - Other (Eye disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes